CLINICAL TRIAL: NCT06507345
Title: Comparative Effectiveness of Opioid Versus Opioid-free Post-discharge Analgesia After Outpatient Breast Surgery: A Protocol for a Randomized Controlled Trial (PAIN-Alt Trial)
Brief Title: Postoperative Analgesia Intervention With Non-opioid Alternatives (PAIN-Alt) Trial - Breast Surgery
Acronym: PAIN-Alt
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Julio F Fiore Jr, Associate Professor, Scientist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-10253
Record Dates: First submitted 2024-07-04; First posted 2024-07-18 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Post Operative Pain; Opioid Analgesic Adverse Reaction; Surgery; Postoperative Pain; Breast Disease
Keywords: Surgery; Postoperative analgesia; Breast surgery; Opioids; Postoperative pain; Postoperative care
MeSH Terms: conditions — Pain, Postoperative; Breast Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Opioid Analgesia (OA) (Active Comparator)
  Interventions: Other: Opioid Analgesia (OA) [Multimodal analgesia including opioid drugs]
- Opioid-Free Analgesia (OFA) (Experimental)
  Interventions: Other: Opioid-Free Analgesia (OFA) [Multimodal analgesia not including opioid drugs]

INTERVENTIONS:
Other: Opioid Analgesia (OA) [Multimodal analgesia including opioid drugs] — In line with current standard care, discharge prescriptions for this group will include around-the-clock non-opioid analgesics (acetaminophen and/or NSAIDs given at regularly scheduled intervals) and opioid tablets 'as needed' for breakthrough pain (i.e., pain that erupts while patients are already taking analgesics). Non-pharmacological pain interventions (i.e., icepacks, music, meditation.) may be recommended by some surgeons as part of standard practice. Given the pragmatic nature of the trial, the specific around-the-clock analgesia and rescue opioid regimens and other non-pharmacological interventions will be determined by the patient's surgeon discretion considering the breast procedure undertaken, co-morbidities, and patient preference.
  Arms: Opioid Analgesia (OA)
Other: Opioid-Free Analgesia (OFA) [Multimodal analgesia not including opioid drugs] — Discharge prescriptions for this group will include around-the-clock non-opioid analgesics (acetaminophen and/or NSAIDs). In case of breakthrough pain, rescue analgesia may be provided by (1) using evidence-based non-pharmacological pain interventions (i.e., icepacks, music, and meditation), (2) adding non-opioid drugs not included in the initial regimen, or (3) switching drugs targeting individual variances in analgesia response. The specific around-the-clock and rescue OFA regimens will be determined by the patient's surgeon considering the type of procedure, co-morbidities, and patient preference.
  Arms: Opioid-Free Analgesia (OFA)

SUMMARY:
North America is experiencing a crisis of opioid use and abuse, partially caused by excessive prescribing by doctors. People often receive their first opioid prescription for pain treatment after outpatient breast surgery (i.e., surgery to remove all or parts of the breast(s), where patients leave the hospital the same day). Many patients misuse these drugs and become addicted. Additionally, many of the opioid pills prescribed to patients are left unused and may be misused by family members, friends, or other community members. To prevent this problem, surgeons can avoid prescribing opioids by prioritizing opioid-free analgesia (i.e., pain treatment using only non-opioid interventions). Prescribing only non-opioid pain medications after surgery is very common in many countries outside of North America; however, few studies have assessed whether opioid-free analgesia is as effective as opioid analgesia after breast surgery. Therefore, the main question driving this study is: For patients who undergo outpatient breast surgery, is pain treatment without opioids as good as pain treatment with opioids?

The proposed trial will compare two groups of patients: one group will receive opioids to treat pain after surgery, while the other group will receive only non-opioid medications. The impact of these different medication strategies will be measured on pain intensity, pain interference with daily activities, medication side effects, and other outcomes. An expert team of scientists, surgeons, pain specialists, nurses, and patients has been assembled to maximize the success of this study. The results will provide important information to guide surgeons' decisions to prescribe (or not to prescribe) opioids. If opioid-free analgesia is found to be effective, doctors may be able to substantially reduce opioid prescribing after breast surgery and prevent more people from misusing opioids.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing mastectomy (i.e., total, modified radical, radical, or skin/nipple sparing) or lumpectomy (i.e., excisional biopsy, partial or segmental mastectomy, oncoplastic breast-conserving surgery) for malignant (cancer) and non-malignant diseases (i.e., ductal carcinoma in situ)
* Planned discharge on the day of the operation.

Exclusion Criteria:

* Immediate breast reconstruction, i.e., implant, tissue-expander, or autologous/flap-based (often leads to higher levels of pain and analgesia requirements)
* Contraindications to the drugs used in the trial in accordance with Health Canada Monographs (i.e., opioid use disorder, pregnancy, breastfeeding, heart failure, allergy/hypersensitivity, peptic ulcer, bleeding disorders, renal or liver impairment)
* Taking opioids preoperatively
* Cognitive impairment precluding patient-reported outcome assessment
* Need for postoperative hospitalization decided before randomization (i.e., same-day discharge cancelled for medical [e.g., intra-operative complications] or non-medical reasons [e.g., lack of support at home]).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Postoperative days 1 to 7.
  Pain intensity will be measured using the Brief Pain Inventory-Short Form (BPI), a self-reported pain questionnaire developed by the World Health Organization (WHO). In this questionnaire, pain intensity is measured across four domains (worst, least, on average, and currently). Aggregated scores of pain intensity range from 0-10, with higher scores representing worse outcomes.
Pain interference | Postoperative days 1 to 7.
  Pain interference will be measured using the Brief Pain Inventory-Short Form (BPI), a self-reported pain questionnaire developed by the World Health Organization (WHO). In this questionnaire, pain interference is measured across seven domains (mood, work, general activity, walking, relationships, enjoyment of life, and sleep). Aggregated scores of pain interference range from 0-10, with higher scores representing worse outcomes.

SECONDARY OUTCOMES:
Adverse drug events | Up to 30 days after surgery.
  Data regarding adverse drug events will be obtained from an author-generated questionnaire and from medical records.
  Adverse events will be coded using the MedDRA coding dictionary, grade their severity according to the Common Terminology Criteria for Adverse Events (CTCAE) (1-Mild to 5-Death) and assess potential causality using the WHO/UMC system (certain, probable/likely, possible, unlikely, conditional/unclassified, or un-assessable/un-classifiable).
Time to stopping pain medication | Up to 30 days after surgery.
  The time to the first report of stopping the use of pain medication will be calculated based on information obtained via questionnaires responded on day 1 to 7, and weeks 2, 3 and 4 after surgery. The time to stopping pain medication will be calculated based on the first of two consecutive reports of 'no pain medication'.
Physical and Mental Health Status | Postoperative weeks 1, 2, 3, and 4, postoperative month 3 and 6.
  This outcome will be assessed using PROMIS-29, a generic health survey, which assesses 8 domains of health (physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social roles and activities, pain interference, and pain intensity).
Opioid misuse | Postoperative weeks 1, 2, 3, and 4, postoperative month 3 and 6.
  This outcome will be assessed using Prescription Opioid Misuse Index which is a 6-item questionnaire includes questions regarding excessive dose, frequency of use, need for early refills, feeling high from the medication, taking the medication due to stress and obtaining prescriptions from multiple physicians.
Satisfaction with pain management | Postoperative day 7.
  Patients will be asked to rate their overall satisfaction with the pain treatment received after discharge using a question adapted from the American Pain Society Patient Outcome Questionnaire: Please rate your satisfaction with the pain treatment that you received since hospital discharge (Scale 0-10; Extremely Dissatisfied-Extremely Satisfied).
30-day postoperative complications | Up to 30 days after surgery.
  Data regarding postoperative complications will be obtained from medical records and graded by severity using the Dindo-Clavien classification. This system grades complications according to the therapy needed for treatment (grades I to IV, best to worse). Complications within 30 days after surgery will be recorded. In addition, the Comprehensive Complication Index (CCI) will be generated for each patient to summarize the complete spectrum of postoperative complications and their severity in a single score ranging from 0 to 100 (best to worse).
30-day unplanned healthcare utilization | Up to 30 days after surgery.
  Unplanned healthcare utilization (ED visits and unplanned hospital readmissions) within 30 days after surgery will be extracted from the electronic medical records and patient self-report.
Chronic postsurgical pain | Up to 6 months after surgery.
  Chronic postsurgical pain will be defined according to ICD-11 as 'pain that develops after a surgical procedure and persists at least 3 months after surgery'. Patients will be asked about chronic pain at 3 and 6 months after surgery using a question modified from the International Pain Outcomes (IPO) Questionnaire. To have a baseline comparator, a similar question will be asked to inquire about the presence of chronic pain preoperatively.
Persistent opioid use | Up to 6 months after surgery.
  The filling of opioid prescriptions will be monitored for 6 months. According to previous literature, persistent opioid use will be defined when a patient has an opioid prescription filled between 90 and 180 days after surgery. Data is obtained via provincial pharmacy records.

CONTACTS AND LOCATIONS:
Overall Officials: Julio Flavio Fiore, PhD, Principal Investigator — McGill University
Locations (1):
- McGill University Health Centre (Glen Site), Montreal, Quebec, Canada

REFERENCES:
- [Background] Fiore JF Jr, El-Kefraoui C, Chay MA, Nguyen-Powanda P, Do U, Olleik G, Rajabiyazdi F, Kouyoumdjian A, Derksen A, Landry T, Amar-Zifkin A, Bergeron A, Ramanakumar AV, Martel M, Lee L, Baldini G, Feldman LS. Opioid versus opioid-free analgesia after surgical discharge: a systematic review and meta-analysis of randomised trials. Lancet. 2022 Jun 18;399(10343):2280-2293. doi: 10.1016/S0140-6736(22)00582-7. PMID 35717988
- [Background] Fiore JF Jr, Olleik G, El-Kefraoui C, Verdolin B, Kouyoumdjian A, Alldrit A, Figueiredo AG, Valanci S, Marquez-GdeV JA, Schulz M, Moldoveanu D, Nguyen-Powanda P, Best G, Banks A, Landry T, Pecorelli N, Baldini G, Feldman LS. Preventing opioid prescription after major surgery: a scoping review of opioid-free analgesia. Br J Anaesth. 2019 Nov;123(5):627-636. doi: 10.1016/j.bja.2019.08.014. Epub 2019 Sep 25. PMID 31563269
- [Background] Do U, El-Kefraoui C, Pook M, Balvardi S, Barone N, Nguyen-Powanda P, Lee L, Baldini G, Feldman LS, Fiore JF Jr; McGill Better Opioid Prescribing Collaboration; Alhashemi M, Antoun A, Barkun JS, Brecht KM, Chaudhury PK, Deckelbaum D, Di Lena E, Dumitra S, Elhaj H, Fata P, Fleiszer D, Fried GM, Grushka J, Kaneva P, Khwaja K, Lapointe-Gagner M, McKendy KM, Meguerditchian AN, Meterissian SH, Montgomery H, Rajabiyazdi F, Safa N, Touma N, Tremblay F. Feasibility of Prospectively Comparing Opioid Analgesia With Opioid-Free Analgesia After Outpatient General Surgery: A Pilot Randomized Clinical Trial. JAMA Netw Open. 2022 Jul 1;5(7):e2221430. doi: 10.1001/jamanetworkopen.2022.21430. PMID 35849399
- [Background] Do U, Pook M, Najafi T, Rajabiyazdi F, El-Kefraoui C, Balvardi S, Barone N, Elhaj H, Nguyen-Powanda P, Lee L, Baldini G, Feldman LS, Fiore JF; McGill Better Opioid Prescribing (MBOP) Collaboration. S110-Opioid-free analgesia after outpatient general surgery: A qualitative study focused on the perspectives of patients and clinicians involved in a pilot trial. Surg Endosc. 2023 Mar;37(3):2269-2280. doi: 10.1007/s00464-022-09472-8. Epub 2022 Aug 2. PMID 35918552
- [Derived] Fiore JF Jr, Shirzadi S, Roversi K, Prakash I, Wong S, Meterissian S, Meguerditchian AN, Desbiens C, Rivard J, Delisle M, Findlay-Shirras L, Abou Khalil J, Maciver A, Quan ML, Verreault K, Johnston S, Feldman L, McDonald EG; Postoperative Analgesia Intervention with Non-opioid Alternatives (PAIN-Alt) Collaboration. Comparative effectiveness of opioid versus opioid-free analgesia after outpatient breast surgery: PAIN-Alt trial protocol. BMJ Open. 2025 Nov 4;15(11):e107258. doi: 10.1136/bmjopen-2025-107258. PMID 41193191